CLINICAL TRIAL: NCT02726022
Title: A Quality of Life Study of PEGASYS® (Peginterferon-Alfa2a) in Combination With COPEGUS® (Ribavirin) in Patients With Chronic Hepatitis C and Persistently Normal ALT Levels
Brief Title: A Quality of Life Study of Peginterferon-Alfa-2a Plus Ribavirin in Participants With Chronic Hepatitis C and Persistently Normal Alanine Transaminase (ALT) Levels
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML20151
Record Dates: First submitted 2016-03-29; First posted 2016-04-01 (Estimated); Results first posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-04

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Chronic Hepatitis C Participants: Participants with chronic hepatitis C, who were under treatment with peg-interferon alfa-2a and ribavirin for four weeks, will be observed up to 24 weeks after end of treatment (EOT) (up to 72 weeks). Peg-interferon alfa-2a and ribavirin will be administered as per treating physician discretion and according to summary of product characteristics.
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Peginterferon alfa-2a — As per treating physician discretion and according to summary of product characteristics.
  Other Names: Pegasys
Drug: Ribavirin — As per treating physician discretion and according to summary of product characteristics.
  Other Names: Copegus

SUMMARY:
Participants with Chronic Hepatitis C (CHC) and normal ALT, who have been under treatment with peginterferon alfa-2a and ribavirin for at least 4 weeks, will be enrolled into this non-interventional, open-label study. The primary aim is to evaluate quality of life according to the 36-Item Short-Form Health Survey (SF-36) questionnaire, modified for the Greek population.

ELIGIBILITY:
Inclusion Criteria:

* Serological confirmation of chronic infection by anti-hepatitis C virus (HCV) assay
* HCV ribonucleic acid (RNA) positive
* CHC with normal transaminases
* Compensated liver disease
* Non-pregnant and willing to use two contraceptive methods (if fertile)
* At least 4 weeks of prior treatment with peginterferon alfa-2a and ribavirin

Exclusion Criteria:

* Pregnant or lactating women
* Co-infection with hepatitis A or B, or human immunodeficiency virus (HIV)
* History of seizures or depression
* History of autoimmune disease, severe heart or lung disease, or renal failure with reduced creatinine clearance
* Uncontrolled thyroid disease
* Severe retinopathy
* Leukopenia or thrombocytopenia
* Bleeding esophageal varices or other evidence of hepatic decompensation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with CHC and persistently normal ALT levels who have been receiving peginterferon alfa-2a and ribavirin for at least 4 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2007-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- Greece (5):
  - Aigaleo - Attiki
  - Athens
  - Heraklion
  - Piraeus
  - Thessaloniki

RESULTS

PARTICIPANT FLOW:
Groups:
- Chronic Hepatitis C Participants: Participants with chronic hepatitis C, who were under treatment with peg-interferon alfa-2a (Pegasys) and ribavirin (Copegus) for four weeks, were observed up to 24 weeks after end of treatment (EOT) (up to 72 weeks). Peg-interferon alfa-2a and ribavirin were administered as per treating physician discretion and according to summary of product characteristics.
Period: Overall Study
Arm/Group | Chronic Hepatitis C Participants
Started | 114
Completed | 78
Not Completed | 36
Not completed — Adverse Event | 14
Not completed — Treatment Failure | 8
Not completed — Poor Compliance | 13
Not completed — Treatment Failure and Poor Compliance | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all enrolled participants.
Groups:
- Chronic Hepatitis C Participants: Participants with chronic hepatitis C, who were under treatment with peg-interferon alfa-2a and ribavirin for four weeks, were observed up to 24 weeks after EOT (up to 72 weeks). Peg-interferon alfa-2a and ribavirin were administered as per treating physician discretion and according to summary of product characteristics.
Arm/Group | Chronic Hepatitis C Participants
Number analyzed (Participants) | 114
Age, Continuous [Mean (Standard Deviation); unit: years] — Number of participants analyzed for age were 113.
  years | 46.30 (13.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 59

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) General Health Domain at End of Treatment (EOT)
Description: SF-36 is a standardized survey evaluating 8 domains of functional health and wellbeing: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for general health domain was an average of the individual question scores of this domain, which are scaled 0-100 (100=highest level of functioning). Data was reported by status of gender (male and female) and drug addiction (yes and no).
Time Frame: Baseline, EOT (up to 48 weeks)
Population: Analysis population included all enrolled participants. Number of participants analyzed = participants with evaluable data. Participants evaluable for Gender = 76; participants evaluable for Drug Addiction = 75. Same participants could be evaluated under Gender and Drug Addiction.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chronic Hepatitis C Participants
Number analyzed (Participants) | 76
units on a scale
  Gender: Male | -3.2 (24.6)
  Gender: Female | -3.0 (29.2)
  Drug Addiction: Yes | -7.4 (26.5)
  Drug Addiction: No | -1.2 (27.1)
Statistical Analysis 1: Comparison: Chronic Hepatitis C Participants; The statistical significance of change from baseline to EOT between gender status (male vs female) was tested using Fisher's exact test; Test type: Superiority or Other; p = 0.647, Fisher Exact
Statistical Analysis 2: Comparison: Chronic Hepatitis C Participants; The statistical significance of change from baseline to EOT between drug addiction status (yes vs no) was tested using Fisher's exact test; Test type: Superiority or Other; p = 0.373, Fisher Exact

2. Primary Outcome: Change From Baseline in SF-36 General Health Domain at 24 Weeks After EOT
Description: as for outcome 1
Time Frame: Baseline, 24 weeks after EOT (up to 72 weeks)
Population: Analysis population included all enrolled participants. Number of participants analyzed = participants with evaluable data. Participants evaluable for Gender = 56; participants evaluable for Drug Addiction = 56. Same participants could be evaluated under Gender and Drug Addiction.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chronic Hepatitis C Participants
Number analyzed (Participants) | 56
units on a scale
  Gender: Male | 0.3 (26.3)
  Gender: Female | 15.4 (25.0)
  Drug Addiction: Yes | 8.4 (18.7)
  Drug Addiction: No | 7.6 (29.1)
Statistical Analysis 1: Comparison: Chronic Hepatitis C Participants; The statistical significance of change from baseline to 24 weeks after EOT between gender status (male vs female) was tested using Fisher's exact test; Test type: Superiority or Other; p = 0.049, Fisher Exact
Statistical Analysis 2: Comparison: Chronic Hepatitis C Participants; The statistical significance of change from baseline to 24 weeks after EOT between drug addiction status (yes vs no) was tested using Fisher's exact test; Test type: Superiority or Other; p = 0.860, Fisher Exact

3. Primary Outcome: Change From Baseline in SF-36 Physical Component Summary (PCS) at EOT
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and wellbeing: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a domain was an average of the individual question scores, which were scaled 0-100 (100=highest level of functioning). Score from physical function, role physical, bodily pain, and general health domains were averaged to calculate PCS. Total score range for PCS was 0-100 (100=highest level of physical functioning).
Time Frame: Baseline, EOT (up to 48 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chronic Hepatitis C Participants
Number analyzed (Participants) | 76
units on a scale
  Gender: Male | -0.7 (24.6)
  Gender: Female | 0.17 (26.5)
  Drug Addiction: Yes | -0.4 (18.7)
  Drug Addiction: No | -0.1 (27.7)
Statistical Analysis 1: Comparison: Chronic Hepatitis C Participants; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.921, Fisher Exact
Statistical Analysis 2: Comparison: Chronic Hepatitis C Participants; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.962, Fisher Exact

4. Primary Outcome: Change From Baseline in SF-36 PCS at 24 Weeks After EOT
Description: as for outcome 3
Time Frame: Baseline, 24 weeks after EOT (up to 72 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chronic Hepatitis C Participants
Number analyzed (Participants) | 56
units on a scale
  Gender: Male | 0.1 (27.5)
  Gender: Female | 15.8 (23.8)
  Drug Addiction: Yes | 6.7 (17.1)
  Drug Addiction: No | 8.4 (29.6)
Statistical Analysis 1: Comparison: Chronic Hepatitis C Participants; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.052, Fisher Exact
Statistical Analysis 2: Comparison: Chronic Hepatitis C Participants; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.677, Fisher Exact

5. Primary Outcome: Change From Baseline in SF-36 Mental Component Summary (MCS) at EOT
Description: SF-36 is a standardized survey evaluating 8 domains of functional health and wellbeing: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a domain was an average of the individual question scores, which were scaled 0-100 (100=highest level of functioning). Score from mental health, role emotional, social functioning, and vitality domains were averaged to calculate MCS. Total score range for MCS was 0-100 (100=highest level of mental functioning).
Time Frame: Baseline, EOT (up to 48 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chronic Hepatitis C Participants
Number analyzed (Participants) | 76
units on a scale
  Gender: Male | -5.10 (25.9)
  Gender: Female | -3.47 (25.3)
  Drug Addiction: Yes | -9.4 (23.3)
  Drug Addiction: No | -2.1 (26.2)
Statistical Analysis 1: Comparison: Chronic Hepatitis C Participants; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.720, Fisher Exact
Statistical Analysis 2: Comparison: Chronic Hepatitis C Participants; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.237, Fisher Exact

6. Primary Outcome: Change From Baseline in SF-36 MCS at 24 Weeks After EOT
Description: as for outcome 5
Time Frame: Baseline, 24 weeks after EOT (up to 72 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chronic Hepatitis C Participants
Number analyzed (Participants) | 56
units on a scale
  Gender: Male | -3.2 (27.1)
  Gender: Female | 6.5 (30.7)
  Drug Addiction: Yes | 4.4 (26.4)
  Drug Addiction: No | 0.9 (30.6)
Statistical Analysis 1: Comparison: Chronic Hepatitis C Participants; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.184, Fisher Exact
Statistical Analysis 2: Comparison: Chronic Hepatitis C Participants; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.889, Fisher Exact

ADVERSE EVENTS:
Time Frame: Baseline up to Week 72
Description: Due to observational nature of the study only serious adverse events and peginterferon-alfa 2a-related non-serious adverse event were collected.
Arm/Group | Chronic Hepatitis C Participants
Serious Adverse Events (participants affected / at risk) | 1/114
Other Adverse Events (participants affected / at risk) | 27/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chronic Hepatitis C Participants (N=114)
Hypertensive Crisis (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chronic Hepatitis C Participants (N=114)
Anemia (Blood and lymphatic system disorders) | 13
Leucopenia (Blood and lymphatic system disorders) | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 6
Fatigue (General disorders) | 8
Fever (General disorders) | 6
Headache (General disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.